CLINICAL TRIAL: NCT07366424
Title: Evaluating the Impact of "CHUT OTONOM®" Footwear on the Spatio-temporal Parameters of Walking and the Risk of Falls in Elderly People at High Risk of Falling.
Acronym: CHAUSS-THERA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: INNOTHERA Laboratories (Unknown); SEED at Lille University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024_0604
Record Dates: First submitted 2025-12-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Falls in the Elderly
Keywords: Fall, elderly, balance, walking, therapeutic footwear, CHUT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: "CHUT OTONOM®" shoes from Innothera Laboratories (Experimental): Once the patient has agreed to participate, they will be asked to put on, depending on their randomization arm (sequence):
  Sequence 1: "CHUT OTONOM®" shoes from Innothera Laboratories to perform the TUG, the one-leg stand test, and the treadmill recording (GaitRite) for 5 minutes. After a 15-minute rest period, the measurements will then be taken with their usual shoes.
  Interventions: Device: "CHUT OTONOM®" shoes from Innothera Laboratories
- Sequence 2: Their usual shoes to perform the TUG (Active Comparator): Once the patient has agreed to participate, they will be asked to put on, depending on their randomization arm (sequence):
  Sequence 2: Their usual shoes to perform the TUG, the one-leg stand test, and the treadmill recording (GaitRite) for 5 minutes. After a 15-minute rest period, the measurements will then be taken with the "CHUT OTONOM®" shoes from Innothera Laboratories
  Interventions: Device: "CHUT OTONOM®" shoes from Innothera Laboratories

INTERVENTIONS:
Device: "CHUT OTONOM®" shoes from Innothera Laboratories — The patient will be asked to put on, depending on the group to which they have been randomized, Sequence 1: "CHUT OTONOM®" shoes from Innothera Laboratories to perform the Timed Up and Go (TUG) test, the one-leg balance test, and the treadmill recording (GaitRite) for 5 minutes. After a 15-minute rest period, the same measurements will then be taken with their usual shoes.
  Arms: Sequence 1: "CHUT OTONOM®" shoes from Innothera Laboratories
Device: "CHUT OTONOM®" shoes from Innothera Laboratories — The patient will be asked to put on, depending on the group to which they have been randomized, Sequence 2: "Their usual shoes to perform the TUG, the one-leg stand test, and the treadmill recording (GaitRite) for 5 minutes. After a 15-minute rest period, the same measurements will then be taken with the "CHUT OTONOM®" shoes from Innothera Laboratories
  Arms: Sequence 2: Their usual shoes to perform the TUG

SUMMARY:
Footwear is one of the extrinsic factors that can cause falls in older adults. Indeed, ill-fitting or worn shoes or slippers that do not support the foot properly, have slippery soles or high heels can contribute to falls. The quality of footwear is a modifiable risk factor that must be addressed to reduce the risk of falling. Therefore, examining the feet and assessing footwear are an integral part of the clinical evaluation of older adults at risk of falling, Older patients are advised to wear shoes and to limit the use of slippers or slipper socks, which do not provide adequate support for the feet and may increase the risk of falls.

In this regard, in November 2020, the French National Authority for Health (HAS) published best practice recommendations entitled "The feet of older people: medical approach and podiatric care." INNOTHERA Laboratories recently designed a new line of shoes, called CHUT OTONOM®, featuring a patented outsole whose effectiveness in terms of stability has been proven in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 65 years of age or older
* Having fallen at least once in the previous 6 months.
* Patients whose foot morphology corresponds to the sizes available in Innothera Laboratories' "CHUT OTONOM®" shoes (feet with increased volume).
* Patients able to walk 10 meters unaided, without technical or human assistance.
* Patients seen at the "Multidisciplinary Fall Assessment" day hospital at Calmette Hospital, Lille University Hospital.
* Patients who have given their consent to participate in the study (written consent form signed).
* Patients affiliated to a social health insurance scheme (beneficiaries or dependents).

Exclusion Criteria:

* Presence of a focal motor deficit in the lower limbs from neurological or orthopedic causes (e.g., hemiplegia resulting from a stroke, limb amputation, etc.).
* Inability to give informed consent
* Persons under legal protection (guardianship, curatorship, judicial protection)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-02-07 (Estimated); Study Completion 2027-02-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of walking speed (cm/s) using the GaitRite device under two conditions: with Innothera Laboratories' CHUT OTONOM® shoes and with the patient's usual shoes. | Duration of each subject's participation: 7 days
  walking speed (centimeters/seconds)

SECONDARY OUTCOMES:
Double support time (seconds) | Duration of each subject's participation: 7 days
  Measuerd using GaitRite
Stride length (centimeters) | Duration of each subject's participation: 7 days
  Measuerd using GaitRite
Stride length variability (percentage) | Duration of each subject's participation: 7 days
  Measuerd using GaitRite
Cycle duration variability (percentage) | Duration of each subject's participation: 7 days
  Measuerd using GaitRite
Gait asymmetry (percentage), | Duration of each subject's participation: 7 days
  Measuerd using GaitRite
Timed Up and Go Test scores in single-task and dual-task conditions. | Duration of each subject's participation: 7 days
  Higher scores mean a worse outcome
Shoe comfort will be evaluated using the following subjective ordinal scale: 1 very uncomfortable, 2 uncomfortable, 3 neutral, 4 comfortable, 5 very comfortable (according to Menant et al., 2008) on D1 and D7. | Duration of each subject's participation: 7 days
  Shoe comfort assessed on a Likert scale from 1 to 5 on Day 1 and Day 7
The ease of putting on and taking off shoes will be evaluated using the following modified subjective ordinal scale (Menant et al., 2008): 1 very difficult, 2 difficult, 3 neutral, 4 easy, 5 very easy on D1 and D7. | Duration of each subject's participation: 7 days
  Ease of putting on and taking off shoes assessed on a Likert scale from 1 to 5 on Day 1 and Day
The feeling of stability will be evaluated using the following subjective ordinal scale (Menant et al., 2008): 1 very unstable, 2 unstable, 3 neutral, 4 stable, 5 very stable on D1 and D7. | Duration of each subject's participation: 7 days
  Feeling of stability assessed on a Likert scale from 1 to 5 on Day 1 and Day 7
The feeling of security will be evaluated using the following subjective ordinal scale (Menant et al., 2008): 1 always, 2 often, 3 sometimes, 4 rarely, 5 never on D1 and D7 | Duration of each subject's participation: 7 days
  Feeling of security assessed on a Likert scale from 1 to 5 on Day 1 and Day7

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Lille, Lille, France